CLINICAL TRIAL: NCT00469989
Title: Randomised Placebo Controlled Study of Effects of Therapeutic Hookworm Infection in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB08A3
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
Keywords: immune system; allergy; hookworm infection; parasite infection; asthma
MeSH Terms: conditions — Asthma; Hypersensitivity; Hookworm Infections; Parasitic Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Infection with hookworm larvae

SUMMARY:
There has been considerable debate over the last 30 years about the interaction between asthma and parasitic infection. It has been suggested that at least part of the reason for the increasing prevalence of asthma in the developed world is a decrease in parasite infections resulting from improved living conditions with economic development. Our previous studies in Ethiopia suggest that hookworm infection may be particularly important in this process.

To establish definitively whether parasites can protect against allergic disease, and specifically asthma, ultimately requires a randomised clinical trial of parasite infection in patients with asthma. We, the researchers at the University of Nottingham, have completed a study in normal volunteers to establish the dose of hookworms necessary to generate infection at the level shown to be protective in population surveys, and shown that infection is well tolerated. In addition, we have recently completed a randomized placebo-controlled clinical trial of hookworm infection in allergic patients with rhinitis which showed that there was no negative effect on bronchial responsiveness during the phase in the lifecycle where the hookworm larvae migrate through the lungs. Consequently, are now proceeding with the definitive randomized placebo-controlled trial of hookworm infection in people with asthma. This study will also provide us with the opportunity to investigate the cellular mechanisms of the effect of hookworm infection on the immune system.

DETAILED DESCRIPTION:
Epidemiological evidence suggests that human hookworm infection is associated with a reduced risk of asthma and allergic disease. This association is potentially important not only to understanding the aetiology of asthma and allergic disease, but also because it suggests that hookworms or their products might be therapeutically effective in these conditions. To test the hypothesis that hookworms protect against asthma ultimately requires a clinical trial.

We have carried out a dose-ranging study to establish the dose of hookworm larvae necessary to generate infection at the intensity shown to be protective in epidemiological studies, with acceptable side effects. We have also completed a randomized controlled clinical trial of hookworm infection in people with allergic rhinoconjunctivitis and have shown that there is no significant change in airway responsiveness during the lung migration phase of the hookworm life cycle. We are now performing the definitive study which is a randomized placebo-controlled trial of the effects of therapeutic hookworm infection in people with asthma. During this study, we will be monitoring various indicators of asthma control but will also be able to measure a range of relevant immunological parameters to explore the relation between these parameters and expression of the allergic and asthmatic phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Use of regular inhaled corticosteroid treatment to a maximum of 1000mcg beclomethasone or equivalent per day
* Measurable airway responsiveness to AMP
* Negative hookworm serology
* Positive skin prick tests to D.pteronyssinum, cat fur or grass pollen

Exclusion Criteria:

* Possible or planned pregnancy or breastfeeding
* Use of regular oral corticosteroids or immunosuppressive medication
* Anemia
* History of anaphylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline airway responsiveness to adenosine-5-monophosphate (AMP) during the 12 weeks of the study.

SECONDARY OUTCOMES:
Change in peak flow variability, asthma symptom scores, asthma medication usage, allergen skin wheal response,total and specific IgE titres, acidic mammalian chitinase, cytokine profiles, other inflammatory markers
occurrence of adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: John Britton, Principal Investigator — University of Nottingham; David Pritchard, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom